CLINICAL TRIAL: NCT01572155
Title: Pilot Study: Anti-inflammatory Effect of Peroperative Stimulation of the Vagus Nerve: Potential New Therapeutic Intervention to Shorten Postoperative Ileus
Brief Title: Pilot Study: Anti-inflammatory Effect of Peroperative Stimulation of the Vagus Nerve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Guy Boeckxstaens, Principal Investigator, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S53497
Record Dates: First submitted 2012-04-02; First posted 2012-04-06 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Postoperative Ileus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sham stimulation (No Intervention): No stimulation of nervus vagus
- Vagus stimulation 1 (Active Comparator): 2 times 2 minutes (beginning and end of surgery) stimulation at 5 Hz, 500 micro s, 2.5 mA
  Interventions: Procedure: Vagus stimulation 1
- Vagus stimulation 2 (Active Comparator): 2 times 2 minutes (beginning and end of surgery) stimulation at 20 Hz, 500 micro s, 2.5 mA
  Interventions: Procedure: Vagus stimulation 2

INTERVENTIONS:
Procedure: Vagus stimulation 1 — 2 times 2 minutes (beginning and end of surgery) stimulation at 5 Hz, 500 micro s, 2.5 mA
  Arms: Vagus stimulation 1
Procedure: Vagus stimulation 2 — 2 times 2 minutes (beginning and end of surgery) stimulation at 20 Hz, 500 micro s, 2.5 mA
  Arms: Vagus stimulation 2

SUMMARY:
Hypothesis:

Electrical stimulation of the abdominal vagus nerve has an anti-inflammatory effect and represents a new therapeutic approach to shorten postoperative ileus.

Aims:

In the present pilot study, the investigators want to evaluate the anti-inflammatory effect of peroperative electrical stimulation of the vagus nerve. To this end, the following aims are formulated:

1. to optimize the technique of intra-operative electrical vagus nerve stimulation
2. to show that electrical stimulation of the intra-abdominal vagus nerve reduces the inflammatory response to abdominal surgery
3. to evaluate whether electrical stimulation of the vagus nerve leads to clinical improvement (collect pilot data)

ELIGIBILITY:
Inclusion Criteria:

* Patients with rectal carcinoma eligible for open rectal resection
* Age between 18 and 70 years

Exclusion Criteria:

* Preoperative therapeutic abdominal radiation
* Evident intra-abdominal inflammation (diagnosed by imaging and/or laboratory test results, including abscess or cholecystitis)
* American Society of Anesthesiologists physical-health status classification (ASA-PS) >3
* Poorly regulated diabetes (>200 mg/dl (=11mmol/l))

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
levels of pro-inflammatory cytokines in serum, peritoneal lavage and supernatant of stimulated PBMCs (peripheral blood mononuclear cell) | From date of surgery until the date of lab analysis (in short time period after taking the blood sample) .Blood samples will be taken before surgery, 2, 24 and 48 hrs after surgery.

SECONDARY OUTCOMES:
gastric stasis (volume of gastric fluid produced by gastric tube on postoperative day 1) | From date of surgery until postoperative day 1.
time to first flatus | From date of surgery until the date of discharge from the hospital.
time to tolerance of oral food intake | From date of surgery until the date of discharge from the hospital
time to tolerance of oral food intake AND first defecation | From date of surgery until the date of discharge from the hospital
gastrointestinal symptoms (nausea, pain, bloating) | From date of surgery until the date of discharge from the hospital
Time to first defecation | From date of surgery until the date of discharge from the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Boeckxstaens, M.D., Principal Investigator — Catholic University Leuven
Locations (1):
- University hospitals Leuven, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Background] Kalff JC, Buchholz BM, Eskandari MK, Hierholzer C, Schraut WH, Simmons RL, Bauer AJ. Biphasic response to gut manipulation and temporal correlation of cellular infiltrates and muscle dysfunction in rat. Surgery. 1999 Sep;126(3):498-509. PMID 10486602
- [Background] Kalff JC, Schraut WH, Simmons RL, Bauer AJ. Surgical manipulation of the gut elicits an intestinal muscularis inflammatory response resulting in postsurgical ileus. Ann Surg. 1998 Nov;228(5):652-63. doi: 10.1097/00000658-199811000-00004. PMID 9833803
- [Derived] Peters EG, De Jonge WJ, Smeets BJ, Luyer MD. The contribution of mast cells to postoperative ileus in experimental and clinical studies. Neurogastroenterol Motil. 2015 Jun;27(6):743-9. doi: 10.1111/nmo.12579. PMID 26011782